CLINICAL TRIAL: NCT02671760
Title: A Randomized, Double-Blind, Single-Dose Study to Assess the Pharmacodynamic Effects of SM-1 Versus Comparator and Placebo in a 5 Hour Phase Advance Model of Insomnia in Adults Who Suffer From Short-Term Insomnia
Brief Title: Pilot Study of a Combination Drug Product for Treatment of Short-term Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sequential Medicine Ltd (Industry)
Collaborators: Clinilabs, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM-A-02
Record Dates: First submitted 2016-01-20; First posted 2016-02-02 (Estimated); Results first posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-01

CONDITIONS: Short-term Insomnia
Keywords: Short-term insomnia; difficulty sleeping; sedative; hypnotic
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment (Experimental): SM-1
  Interventions: Drug: SM-1
- Comparator (Active Comparator): 2-drug combination
  Interventions: Drug: Comparator
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SM-1 — 3-drug combination product containing 50 mg diphenhydramine, 5 mg zolpidem and 0.5 mg lorazepam
  Arms: Treatment
Drug: Comparator — 2-drug combination comprised of 5 mg zolpidem and 0.5 mg lorazepam
  Arms: Comparator
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of a combination drug product containing diphenhydramine, zolpidem and lorazepam on total sleep time. Participants will be adults who sometimes have difficulty falling asleep or staying asleep, but who do not have chronic insomnia. The study involves 3 one-night stays in a sleep center in New York City.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of a combination drug product containing 50 mg diphenhydramine, 5 mg zolpidem and 0.5 mg lorazepam on total sleep time, and to determine the contribution of diphenhydramine to the combination, using a 5-hour Phase Advance model of sleep challenge. This is a 3-arm cross-over study; each participant will receive 3 single-dose treatments on consecutive visits. The 3 arms are: investigational combination product, placebo, and a 2-drug comparator containing the zolpidem and lorazepam components but not diphenhydramine. Participants will be adults who sometimes have difficulty falling asleep or staying asleep, but who are generally healthy and do not have chronic insomnia or sleep apnea.

A total of 39 subjects are being recruited. Subjects who qualify for participation will be asked to keep a sleep diary to document their sleep times leading up to and during the study, and will be asked to spend 7-8 hours in bed at a regular bedtime during the study. Qualifying participants also will not anticipate significant disruptions in their sleep schedules, for example by traveling across timezones or changing shifts at work, during the study. The study requires 3 one-night stays in a sleep center in New York City, for administration of the study treatments and EEG measurements. Qualifying subjects will anticipate being able to return to the sleep center, located in Manhattan, for a total of 4 visits, including initial screening and 3 treatment times.

During each sleep center visit, subjects will be given their study treatment and be put to bed 5 hours before their usual bedtime, and sleep time will be monitored for 8 hours. Each subject will receive all 3 treatments, although the sequence of the 3 treatments will be randomized. Both subjects and study personnel monitoring the subjects will be blinded to the identity of the treatment administered at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 19 and 32 kg/m2, inclusive;
* Report occasional difficulty falling asleep or staying asleep;
* Report a regular, habitual bedtime between 21:00 and 24:00, routinely spend at least 7.5 and no more than 9.0 hours in bed each night and observe a bedtime that does not vary by more than 2 hours over the course of the week. Subjects will be required to complete at least 5 days of sleep information in a diary provided at the screening visit and returned to study personnel no later than 24 hours prior to check-in for the first overnight visit.
* Be in good general health as determined by a thorough medical history and physical examination including vital signs and clinical laboratory tests;
* Females of childbearing potential must be using an acceptable method of contraception, have a negative serum pregnancy test at screening and have a negative urine pregnancy test before randomization and prior to each Treatment Period. Acceptable methods of contraception include oral, intrauterine and injectable contraceptives or double barrier methods. After screening, subjects using oral contraceptives must agree to add a double barrier method until 30 days following the last dose of study medication. Female subjects relying on oral contraceptives must have been using them for at least one month prior to screening;
* Female subjects who have been surgically sterilized are eligible if they have a negative serum pregnancy test at screening and negative urine pregnancy test at check-in for Visits 2 and 3, or are post-menopausal as defined by the cessation of menses for a period of at least 2 years prior to screening or have had a complete hysterectomy;
* Male subjects must use an acceptable method of contraception during the course of the study and for the 30 days following the last dose of study medication. Acceptable methods of contraception include:

  1. Abstinence
  2. A condom and one of the following:

  i. Vasectomy for more than 6 months. ii. Female partner who meets one of the following conditions:
  1. Uses a spermicidal gel or foam; or
  2. Has had a tubal ligation, hysterectomy or bilateral oophorectomy; or
  3. Is post-menopausal (menopause is defined as over the age of 60 years, or between 45 and 60 years being amenorrheic for at least 2 years with plasma follicle stimulating hormone (FSH) level > 30 UI/L); or
* Be able to read, understand, and provide written/dated informed consent before enrolling in the study and must be willing to comply with all study procedures;
* Be willing and able to be confined to the clinical research site for one night in each of 3 treatment periods as required by the protocol.
* Refrain from alcohol on PSG days;
* On the days of check-in for each of the study's two treatment periods, refrain from the use of alcohol and from napping, defined as any sleep episode occurring outside of the subject's main sleep episode of the day;
* Report a recent history of napping of no more than once per week.
* An Epworth Sleepiness Scale score ≤8 at screening.

Exclusion Criteria:

* Clinically significant, acute illness within 14 days prior to screening (Visit 1).
* Clinically significant, unstable medical illness;
* Evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic or neurological disease;
* History of cancer or diabetes;
* A supine blood pressure > 140/90 millimeters mercury (mm/Hg) at screening;
* Heart rate > 100 beats per minute (BPM) at screening;
* Clinically significant psychiatric illness, including chronic psychiatric illness or the history or presence of any Axis I condition;
* History or presence of chronic pain;
* Lifetime history of seizure disorder or serious head injury;
* Clinically significant sleep disorder, including insomnia, sleep apnea, narcolepsy, parasomnia, restless leg syndrome or circadian rhythm disorder;
* Any condition that may affect drug absorption;
* Travel across more than three time zones, an expected change in sleep schedule or involvement in night shift work within one month prior to screening or during the study period;
* Any clinically significant abnormal finding on physical examination, vital signs or clinical laboratory tests, as determined by the Investigator;
* History of allergies, or known sensitivity, hypersensitivity, or adverse reaction to any drug similar to diphenhydramine, zolpidem or lorazepam;
* Pregnant or lactating females;
* Positive serum pregnancy test at Visit 1 or positive urine pregnancy test at check-in for Visit 2 or 3;
* Positive urine drug screen at the Visit 1;
* Recent history (≤ one year) of alcohol or drug abuse, or current evidence of substance dependence or abuse as defined by DSM-V criteria;
* Regular consumption of "large amounts" of xanthine-containing substances (i.e., more than 500 mg of caffeine per day or equivalent amounts of xanthine-containing substances);
* Self-report of a usual consumption of more than 14 units of alcohol per week. One unit of alcohol is equivalent to 12 ounces of beer, 4 ounces of wine or 1 ounce of liquor;
* Use of more than 10 products containing nicotine per day or routinely smokes during sleep period
* Discontinuation of smoking or participation in a smoking cessation program within 90 days of screening;
* Any use with the six months prior to screening of restricted concomitant medications including prescription hypnotics, antidepressants, anxiolytics, anticonvulsants or narcotics;
* Use of any prescription drug, OTC medication, grapefruit juice, herbal preparation or food supplement, excluding vitamins, acetaminophen or hormonal contraceptives within two weeks of randomization;
* Use of any investigational drug within 30 days prior to screening or any prior exposure to the study drugs diphenhydramine, zolpidem or lorazepam or other drugs of the same pharmaceutical classes;
* Positive alcohol breathalyzer test at the time of screening or prior to dosing at Visit 2, 3 or 4.

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dahl, PhD, Study Director — Sequential Medicine Ltd; Maha Ahamad, MD, Principal Investigator — Clinilabs, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dahl T, Chen LB, Zammit G, Ahmad M, Roth T. Efficacy of SM-1 in a transient insomnia model. Hum Psychopharmacol. 2019 Nov;34(6):e2713. doi: 10.1002/hup.2713. PMID 31837050

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: SM-1 Then Comparator Then Placebo: Subjects received a single dose of SM-1 followed by a 5-16 day washout. They the received a single dose of Comparator followed by a 5-16 day washout. They then received a single dose of Placebo.
- Experimental: Comparator Then Placebo Then SM-1: Subjects received a single dose of Comparator followed by a 5-16 day washout. They the received a single dose of Placebo followed by a 5-16 day washout. They then received a single dose of SM-1.
- Experimental: Placebo Then SM-1 Then Comparator: Subjects received a single dose of Placebo followed by a 5-16 day washout. They the received a single dose of SM-1 followed by a 5-16 day washout. They then received a single dose of Comparator.
Period: Overall Study
Arm/Group | Experimental: SM-1 Then Comparator Then Placebo | Experimental: Comparator Then Placebo Then SM-1 | Experimental: Placebo Then SM-1 Then Comparator
Started | 13 | 13 | 13
Completed | 13 | 12 (1 Subject could not be contacted for f/u phone call. Data included in safety and efficacy analyses.) | 13
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants regardless of randomization sequence.
Arm/Group | All Study Participants
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 25
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Total Sleep Time
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment | Comparator | Placebo
Number analyzed (Participants) | 39 | 39 | 39
minutes | 382.9 (57.95) | 339.2 (76.57) | 256.2 (98.15)

2. Secondary Outcome: Latency to Persistent Sleep
Description: Time it takes to fall asleep
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment | Comparator | Placebo
Number analyzed (Participants) | 39 | 39 | 39
minutes | 31.2 (52.34) | 42.1 (52.04) | 50.1 (73.13)

3. Secondary Outcome: Awakenings
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: Awakenings
Arm/Group | Treatment | Comparator | Placebo
Number analyzed (Participants) | 39 | 39 | 39
Awakenings | 12.2 (6.73) | 11.0 (6.61) | 9.6 (5.86)

4. Secondary Outcome: Latency to REM Sleep Onset
Description: Time required to achieve REM sleep
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment | Comparator | Placebo
Number analyzed (Participants) | 39 | 39 | 39
minutes | 112.5 (53.61) | 71.3 (43.89) | 61.2 (36.70)

5. Secondary Outcome: Adverse Events
Description: Safety and tolerability assessed in terms of the incidence of AEs
Time Frame: 8 hours
Measure: Number; unit: Number of Events
Arm/Group | Treatment | Comparator | Placebo
Number analyzed (Participants) | 39 | 39 | 39
Number of Events | 2 | 3 | 2

6. Secondary Outcome: Safety and Tolerability in Terms of Residual Sleepiness
Description: Karolinska Sleepiness Scale. This is a 9-point scale with values ranging from 1 (extremely alert) to 9 (extremely sleepy). Lower scores indicate less residual sleepiness.
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment | Comparator | Placebo
Number analyzed (Participants) | 39 | 39 | 39
Units on a scale | 5.8 (2.06) | 6.0 (1.80) | 6.1 (2.03)

7. Secondary Outcome: Safety and Tolerability in Terms of Residual Sleepiness
Description: Digit Symbol Substitution Test. The test score is number of correct answers in 90 seconds. Higher scores indicate favorable response (i.e., less residual sleepiness). The duration of the challenge is the 90 second time limit; there is no theoretical maximum score to attain.
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: Correct answers
Arm/Group | Treatment | Comparator | Placebo
Number analyzed (Participants) | 39 | 39 | 39
Correct answers | 53.1 (15.97) | 53.3 (13.74) | 55.3 (14.07)

ADVERSE EVENTS:
Time Frame: Entire study, up to 7 days after the last treatment.
Arm/Group | Treatment | Comparator | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 2/39 | 3/39 | 3/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=39) | Comparator (N=39) | Placebo (N=39)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Initial Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No